CLINICAL TRIAL: NCT03402607
Title: Phase II Randomized Trial Comparing Percutaneous Ablation to Hypofractionated Image-Guided Radiation Therapy in Veteran and Non-Veteran, Non-surgical Hepatocellular Carcinoma Patients (PROVE-HCC)
Brief Title: Trial Comparing PLA to HIGRT (PROVE-HCC)
Acronym: PROVE-HCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Duke University (Other)
Collaborators: Durham VA Medical Center (U.S. Federal Agency); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00089525
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Results first posted 2021-12-06 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Unresectable
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Local Ablation (PLA) (Active Comparator): A PLA procedure uses high-energy radio waves to treat liver tumors. Using CT and ultrasound guidance the doctor inserts a thin, needle-like probe into the liver tumor A high-frequency current is then passed through the tip of the probe, which heats the tumor with the goal to destroy the cancer cells. This may be done as an outpatient procedure or a short (1-2 day) hospital stay. PLA is the standard treatment for patients with liver cancer who cannot undergo liver surgery.
  Interventions: Procedure: Percutaneous Local Ablation
- Hypofractionated Image-Guided Radiation Therapy (HIGRT) (Active Comparator): HIGRT is an emerging treatment option for patients with HCC; it utilizes external radiation where multiple beams enter the body from multiple angles to treat the liver cancer over typically 5-10 treatments while minimizing radiation to normal tissues. You will receive between 5-10 fractions (treatments) of radiation. Fraction size will be either 5 or 10 Gy (pronounced Gray, a standard unit of radiation measurement) depending on your tumor size and location or underlying liver function. The total dose of radiation is 50 Gy.
  Interventions: Radiation: Hypofractionated Image Guided Radiation Therapy

INTERVENTIONS:
Procedure: Percutaneous Local Ablation — Microwave Ablation (MWA) is a form of percutaneous localized ablation using thermal ablation techniques to treat cancer via direct coagulative necrosis. Microwaves can generate high temperatures in a short period of time; MWA has the potential to improve treatment efficacy over radiofrequency ablation as it can be used to treat larger lesions and has less susceptibility to heat-sink due to vessel proximity. MWA uses electromagnetic waves (300 MHz to 300 GHz) to produce oscillation of polar molecules within tissue; this generates tissue necrosis through frictional heating. For HCC, one or more microwave antennae are inserted into the liver, usually under the guidance of ultrasonography or computed tomography (CT). Frequency and length of treatment is determined on a case by case basis depending on tumor size and proximity to vessels or other organs at risk.
  Other Names: Microwave Ablation (MWA)
  Arms: Percutaneous Local Ablation (PLA)
Radiation: Hypofractionated Image Guided Radiation Therapy — HIGRT represents the only non-invasive curative modality in the management of HCC. HCC patients typically have a host of other medical comorbidities complicated by underlying liver dysfunction that makes the implementation of liver-directed therapy challenging. Presently HIGRT is typically offered only after alternative surgical (transplantation/hepatectomy) and non-operative approaches (PLA/embolization) have been exhausted.
  Other Names: HIGRT
  Arms: Hypofractionated Image-Guided Radiation Therapy (HIGRT)

SUMMARY:
This phase II, randomized trial compare Quality of Life for patients with Hepatocellular Carcinoma (HCC) who are not surgical candidates or decline surgery and are treated with Percutaneous Local Ablation (PLA) or Hypofractionated Image-Guided Radiation Therapy (HIGRT).

DETAILED DESCRIPTION:
Administrative clarification:

This clinical trial was terminated due to poor enrollment and was replaced by a separate non-randomized trial (NCT04933435).

ELIGIBILITY:
Inclusion Criteria:

* HCC diagnosed either by histology/pathology or Liver Imaging Reporting and Data System (LIRADs 5 per the ACR's LIRADs criteria) by CT or MRI
* Patient is 18 years or older
* ECOG Performance status of 0-2
* Child Pugh score A5, A6, B7 or B8
* Lesions less than or equal to 5cm in size
* Less than or equal to 3 lesions in the liver to be treated on protocol
* Lesion amenable to treatment with both PLA and HIGRT; for PLA treatment this requires the lesion be visible via ultrasound and/or non-contrast CT or feasible per treating physician

Exclusion Criteria:

* Child Pugh score B9 or Class C
* Fluctuating ascites
* Inability to complete baseline QOL forms
* Concurrent administration of systemic therapy for HCC
* Prior liver RT is an exclusion unless subject participation is approved by the PI
* Positive serum pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Palta, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Durham Veterans Administration Medical Center (DVAMC), Durham, North Carolina
  - Duke Cancer Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (7.4) | 65.3 (5.4) | 66.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life (QOL) Using EORTC C-30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30)
Description: To compare change in Quality of Life (QOL), as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC C-30) post treatment in patients receiving PLA vs HIGRT. The EORTC QLQ-C30 reports a Summary Score that is calculated from the mean of 13 of the 15 QLQ-C30 scales (excluding Global Quality of Life scale and the Financial Impact scale). 28 of the items have a range of 1 (not at all) to 4 (very much) and two of them have a range of 1 (very poor) to 7 (excellent). The total summary score ranges from 30 to 126, with lower scores indicating a better quality of life. Only the change in summary score is reported; no individual subscale scores are reported.
Time Frame: Baseline to one month
Population: Participants who completed the EORTC C-30 at both time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 4 | 5
score on a scale | -6.25 [-14.90 to 2.40] | -10.00 [-26.21 to 6.21]

2. Secondary Outcome: Change in Quality of Life (QOL) Using The Functional Assessment of Cancer Therapy - Hepatobiliary (FACT-Hep) Assessment
Description: To compare change in Quality of Life (QOL), as measured by the FACT-Hep questionnaire post treatment in patients receiving PLA vs HIGRT from baseline to 1 month. The FACT-Hep Scale consists of five subscales: Physical well-being (PWB), Social/Family well-being (SWB), Emotional well-being (EWB), Functional well-being (FWB), and the Hepatobiliary Cancer Subscale (HCS). Total score ranges from 0 to 180, with higher scores indicating better quality of life. Average differences in each FACT-Hep Total Score for 3 months minus baseline are reported by treatment arm; no individual subscales are reported. An average difference > 0 indicates improvement in QOL at 3 versus baseline. An average difference < 0 indicates a worsening of QOL at 1 month versus baseline.
Time Frame: Baseline, 1 month, 3 months; change between baseline and 3 months reported
Population: Participants who completed the FACT-Hep at both time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 4 | 5
score on a scale | -14.25 [-39.85 to 11.35] | 0.4 [-34.15 to 33.35]

3. Secondary Outcome: Change in Quality of Life (QOL) Using EORTC QLQ C-30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30)
Description: as for outcome 1
Time Frame: Baseline to 3 months
Population: Participants who completed the EORTC C-30 at both time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 4 | 4
score on a scale | -6.75 [-19.37 to 5.87] | -12.00 [-30.41 to 6.41]

4. Secondary Outcome: Change in Quality of Life (QOL) Using EORTC QLQ C-30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30)
Description: To compare change in Quality of Life (QOL), as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC C-30) post treatment in patients receiving PLA vs HIGRT. To compare change in Quality of Life (QOL), as defined by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC C-30) post treatment in patients receiving PLA vs HIGRT. The EORTC QLQ-C30 reports a Summary Score that is calculated from the mean of 13 of the 15 QLQ-C30 scales (excluding Global Quality of Life scale and the Financial Impact scale). 28 of the items have a range of 1 (not at all) to 4 (very much) and two of them have a range of 1 (very poor) to 7 (excellent). The total summary score ranges from 30 to 126, with lower scores indicating a better quality of life. Only the change in summary score is reported; no individual subscale scores are reported.
Time Frame: Baseline to 6 months
Population: Participants who completed the EORTC C-30 at both time points.
Measure: Mean (95% Confidence Interval); unit: difference in scores on a scale
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 5 | 4
difference in scores on a scale | -11.00 [-26.85 to 4.81] | -9.20 [-30.51 to 12.11]

5. Secondary Outcome: Number of Participants With Grade 2 or Higher Adverse Events
Description: Grade ≥2 acute toxicity within 90 days of treatment initiation for each treatment as defined by the CTCAE v4.0
Time Frame: Up to 90 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 6 | 6
Participants | 1 | 1

6. Secondary Outcome: The Total Healthcare System Costs Associated With PLA vs HIGRT
Description: Healthcare system costs estimated based on national averages for billable charges for all codes associated with PLA vs HIRGT throughout the course of treatment through 90 days post treatment.
Time Frame: From time of intervention to 90 days post treatment
Population: Data not collected.
Arm/Group | Percutaneous Local Ablation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Groups:
- Percutaneous Local Abalation (PLA): A PLA procedure uses high-energy radio waves to treat liver tumors. Using CT and ultrasound guidance the doctor inserts a thin, needle-like probe into the liver tumor A high-frequency current is then passed through the tip of the probe, which heats the tumor with the goal to destroy the cancer cells. This may be done as an outpatient procedure or a short (1-2 day) hospital stay. PLA is the standard treatment for patients with liver cancer who cannot undergo liver surgery.
  Percutaneous Local Ablation: Microwave Ablation (MWA) is a form of percutaneous localized ablation using thermal ablation techniques to treat cancer via direct coagulative necrosis. Microwaves can generate high temperatures in a short period of time; MWA has the potential to improve treatment efficacy over radiofrequency ablation as it can be used to treat larger lesions and has less susceptibility to heat-sink due to vessel proximity. MWA uses electromagnetic waves (300 MHz to 300 GHz) to produce oscillation of polar molecules within tissue; this generates tissue necrosis through frictional heating. For HCC, one or more microwave antennae are inserted into the liver, usually under the guidance of ultrasonography or computed tomography (CT). Frequency and length of treatment is determined on a case by case basis depending on tumor size and proximity to vessels or other organs at risk.
Arm/Group | Percutaneous Local Abalation (PLA) | Hypofractionated Image-Guided Radiation Therapy (HIGRT)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Local Abalation (PLA) (N=6) | Hypofractionated Image-Guided Radiation Therapy (HIGRT) (N=6)
Hospitalization (General disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Local Abalation (PLA) (N=6) | Hypofractionated Image-Guided Radiation Therapy (HIGRT) (N=6)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/07/NCT03402607/Prot_SAP_000.pdf